CLINICAL TRIAL: NCT01572740
Title: A 36-week, Randomised, Multi-centre, Double-blind, Parallel Group Trial to Investigate the Efficacy and Safety of Liraglutide in Combination With Insulin Therapy Compared to Insulin Monotherapy in Japanese Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Liraglutide in Combination With Insulin Therapy Compared to Insulin Alone in Japanese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3925; U1111-1122-4320 (Other: WHO); JapicCTI-121802 (Other: JAPIC)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lira+Insulin (Experimental)
  Interventions: Drug: liraglutide; Drug: insulin
- Placebo+Insulin (Placebo Comparator)
  Interventions: Drug: placebo; Drug: insulin

INTERVENTIONS:
Drug: liraglutide — Liraglutide administered subcutaneously (s.c., under the skin) for 36 weeks combined with insulin therapy.
  Arms: Lira+Insulin
Drug: placebo — Liraglutide placebo administered subcutaneously (s.c., under the skin) for 36 weeks combined with insulin therapy.
  Arms: Placebo+Insulin
Drug: insulin — All subjects will continue their pre-trial insulin therapy (basal, premixed or basal-bolus regimen) during the trial. Insulin dose is fixed for the first 16 weeks and for the subsequent 20 weeks, insulin dose is individually adjusted.

SUMMARY:
This trial is conducted in Asia. The purpose of the trial is to investigate the efficacy and safety of liraglutide in combination with insulin therapy compared to insulin alone in Japanese subjects with type 2 diabetes mellitus. Subjects will remain on their pre-trial insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Current insulin therapy (basal insulin, premixed insulin or basal-bolus regimen) in addition to diet and exercise therapy for at least 12 weeks prior to trial start. Their therapy is stable and fluctuation of total daily insulin dose is within plus/minus 20% for at least 12 weeks prior to trial start and current total daily insulin dose equal to or greater than 10 (I)U/day
* Glycosylated haemoglobin (HbA1c) between 7.5 and 11.0% (both inclusive)
* Body Mass Index (BMI) below 45.0 kg/m^2

Exclusion Criteria:

* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as, but not limited to systemic corticosteroids, beta-antagonists or monoamine oxidase (MAO) inhibitors
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic episode during last 12 months) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Known proliferative retinopathy or maculopathy requiring treatment according to the investigator
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonist within 12 weeks prior to screening
* Treatment with any oral antidiabetic drugs (OADs) within 12 weeks prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2012-04-05 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2013-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (22):
- Japan (22):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi, Kanagawa
  - Novo Nordisk Investigational Site, Ebina-shi
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Katsushika-ku, Tokyo
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokohama

REFERENCES:
- [Result] Seino Y, Kaneko S, Fukuda S, Osonoi T, Shiraiwa T, Nishijima K, Bosch-Traberg H, Kaku K. Combination therapy with liraglutide and insulin in Japanese patients with type 2 diabetes: A 36-week, randomized, double-blind, parallel-group trial. J Diabetes Investig. 2016 Jul;7(4):565-73. doi: 10.1111/jdi.12457. Epub 2016 Jan 23. PMID 27182042
- [Result] Kaneko S, Nishijima K, Bosch-Traberg H, Kaku K, Seino Y. Efficacy and safety of adding liraglutide to existing insulin regimens in Japanese patients with type 2 diabetes mellitus: A post-hoc analysis of a phase 3 randomized clinical trial. J Diabetes Investig. 2018 Jul;9(4):840-849. doi: 10.1111/jdi.12793. Epub 2018 Feb 5. PMID 29277968
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 23 sites in Japan.
Pre-assignment Details: Subjects on pre-trial insulin (basal insulin [intermediate acting human insulin, intermediate acting insulin analogue or long-acting insulin analogue], premixed insulin or basal-bolus regimen) therapy for at least 12 weeks prior to screening.
Groups:
- Lira + Insulin: Liraglutide was administered subcutaneously (s.c., under the skin) once daily (OD) for 36 weeks combined with insulin therapy. The starting dose of the liraglutide was 0.3 mg (50 μL)/day; dose was escalated to 0.6 mg (100 μL)/day and 0.9 mg (150 μL)/day during first 2 weeks; dose was maintained at 0.9 mg (150 μL)/day for subsequent 34 weeks.
  All subjects continued their pre-trial insulin therapy (basal: once daily [OD] or twice daily [BID], premixed: OD or BID or basal-bolus regimen [basal: OD or BID and bolus: three times a day]). Insulin dose was not changed for any subject for the first 16 weeks and for the subsequent 20 weeks, insulin dose was individually adjusted.
- Placebo + Insulin: Liraglutide placebo was administered subcutaneously (s.c., under the skin) OD for 36 weeks combined with insulin therapy. The starting dose of the placebo was 50 μL/day; dose was escalated to100 μL/day and 150 μL/day during first 2 weeks; dose was maintained at 150 μL/day for subsequent 34 weeks.
  All subjects continued their pre-trial insulin therapy (basal: once daily [OD] or twice daily [BID], premixed: OD or BID or basal-bolus regimen [basal: OD or BID and bolus: three times a day]). Insulin dose was not changed for any subject for the first 16 weeks and for the subsequent 20 weeks, insulin dose was individually adjusted.
Period: Overall Study
Arm/Group | Lira + Insulin | Placebo + Insulin
Started | 127 | 130
Completed | 121 | 125
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — unclassified | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira + Insulin | Placebo + Insulin | Total
Number analyzed (Participants) | 127 | 130 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.0) | 59.8 (11.3) | 60.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 113
  Male | 69 | 75 | 144
Body Weight [Mean (Standard Deviation); unit: kg] | 67.7 (15.2) | 65.9 (13.0) | 66.8 (14.1)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.51 (2.42) | 8.79 (2.51) | 8.65 (2.47)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.8 (0.9) | 8.8 (0.9) | 8.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 16
Description: Estimated mean change from baseline in HbA1c after 16 Weeks of treatment.
Time Frame: Week 0, Week 16
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products. Missing data were imputed using last observation carried forward (LOCF). 1 subject in the placebo group did not contribute to the statistical analysis at Week 16 as subject was withdrawn from the trial before sampling for any efficacy data.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
percentage of glycosylated haemoglobin | -1.73 (0.06) | -0.43 (0.06)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimated treatment difference, Mean = -1.30, 95% CI [-1.47 to -1.13]

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 36
Description: Estimated mean change from baseline in HbA1c after 36 Weeks of treatment
Time Frame: Week 0, Week 36
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products. Missing data were imputed using last observation carried forward (LOCF). 1 subject in the placebo group did not contribute to the statistical analysis at Week 36 as subject was withdrawn from the trial before sampling for any efficacy data.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
percentage of glycosylated haemoglobin | -1.68 (0.06) | -0.88 (0.06)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimated treatment difference, Mean = -0.81, 95% CI [-0.99 to -0.63]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 16
Description: Estimated mean change from baseline in FPG after 16 Weeks of treatment.
Time Frame: Week 0, Week 16
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
mmol/L | -1.31 (0.17) | -0.48 (0.17)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p < 0.0006, ANCOVA; Estimated treatment difference, Mean = -0.83, 95% CI [-1.30 to -0.36]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 36
Description: Estimated mean change from baseline in FPG after 36 Weeks of treatment.
Time Frame: Week 0, Week 36
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
mmol/L | -1.55 (0.16) | -1.29 (0.16)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.2511, ANCOVA; Estimated treatment difference, Mean = -0.26, 95% CI [-0.70 to 0.18]

5. Secondary Outcome: Change in Mean Plasma Glucose (PG) of 7-Point Profile From Baseline to Week 16
Description: Estimated mean change from baseline in mean PG of 7-point profile (7-points were before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner and at bedtime) after 16 Weeks of treatment.
Time Frame: Week 0, Week 16
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products. Missing data were imputed using last observation carried forward (LOCF). 9 subjects did not contribute to the statistical analysis at Week 16 due to missing data.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 124 | 124
mmol/L | -2.41 (0.18) | -0.53 (0.18)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimated treatment difference, Mean = -1.87, 95% CI [-2.37 to -1.38]

6. Secondary Outcome: Change in Mean Plasma Glucose (PG) of 7-Point Profile From Baseline to Week 36
Description: Estimated mean change from baseline in mean PG of 7-point profile (7-points were before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner and at bedtime) after 36 Weeks of treatment.
Time Frame: Week 0, Week 36
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products. Missing data were imputed using last observation carried forward (LOCF). 8 subjects did not contribute to the statistical analysis at Week 36 due to missing data.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 124 | 125
mmol/L | -2.65 (0.16) | -1.37 (0.16)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimated treatment difference, Mean = -1.28, 95% CI [-1.73 to -0.83]

7. Secondary Outcome: Change in Mean Prandial PG Increment of 7-Point Profile From Baseline to Week 16
Description: Estimated mean change from baseline in mean prandial PG increment of 7-point profile (7-points were before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner and at bedtime) after 16 Weeks of treatment.
Time Frame: Week 0, Week 16
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 124 | 124
mmol/L | -1.34 (0.17) | -0.61 (0.17)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.0023, ANCOVA; Estimated treatment difference, Mean = -0.73, 95% CI [-1.20 to -0.26]

8. Secondary Outcome: Change in Mean Prandial PG Increment of 7-Point Profile From Baseline to Week 36
Description: Estimated mean change from baseline in mean prandial PG increment of 7-point profile (7-points were before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner and at bedtime) after 36 Weeks of treatment.
Time Frame: Week 0, Week 36
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products. Missing data were imputed using last observation carried forward (LOCF). 13 subjects did not contribute to the statistical analysis at Week 36 due to missing data.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 122 | 122
mmol/L | -1.34 (0.21) | -0.94 (0.21)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.1787, ANCOVA; Estimated treatment difference, Mean = -0.39, 95% CI [-0.97 to 0.18]

9. Secondary Outcome: Change in Body Weight From Baseline to Week 16
Description: Estimated mean change in body weight after 16 Weeks of treatment
Time Frame: Week 0, Week 16
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
kg | -0.42 (0.14) | -0.28 (0.14)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.4806, ANCOVA; Estimated treatment difference, Mean = -0.14, 95% CI [-0.54 to 0.25]

10. Secondary Outcome: Change in Body Weight From Baseline to Week 36
Description: Estimated mean change in body weight after 36 Weeks of treatment
Time Frame: Week 0, Week 36
Population: as for outcome 2
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 129
kg | 0.17 (0.20) | 0.52 (0.20)
Statistical Analysis 1: Comparison: Lira + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.2074, ANCOVA; Estimated treatment difference, Mean = -0.35, 95% CI [-0.91 to 0.20]

11. Secondary Outcome: Number of Adverse Events (AEs)
Description: An AE was defined as treatment emergent if the onset date was on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Week 0 to Week 36 (inclusive)
Population: Safety analysis set includes all subjects who received at least one dose of the trial products.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 130
Events/100 years of patient exposure
  Adverse Events | 449 | 350
  Serious Adverse Events | 8 | 5
  Severe Adverse Events | 5 | 1
  Moderate Adverse Events | 8 | 14
  Mild Adverse Events | 436 | 335

12. Secondary Outcome: Number of Confirmed Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and until the last day on randomised treatment. Confirmed hypoglycaemic episode was defined as hypoglycaemic episodes categorised to severe and/or minor hypoglycaemic episodes.
  Confirmed hypoglycaemia: subject unable to treat himself/herself and/or have a recorded PG < 3.1 mmol/L (56 mg/dL). Minor: PG < 3.1 mmol/L (56 mg/dL).
Time Frame: Week 0 to week 36 (inclusive)
Population: Safety analysis set includes all subjects who received at least one dose of the trial products.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | Lira + Insulin | Placebo + Insulin
Number analyzed (Participants) | 127 | 130
Episodes/100 years of patient exposure | 146 | 187

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a timeframe of 36 weeks + 7 days follow up.
Description: Safety analysis set includes all subjects who received at least one dose of the trial products.
Arm/Group | Lira + Insulin | Placebo + Insulin
Serious Adverse Events (participants affected / at risk) | 6/127 | 4/130
Other Adverse Events (participants affected / at risk) | 93/127 | 69/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira + Insulin (N=127) | Placebo + Insulin (N=130)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain stem thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira + Insulin (N=127) | Placebo + Insulin (N=130)
Diabetic retinopathy (Eye disorders) | 9 (9) | 13 (16)
Constipation (Gastrointestinal disorders) | 15 (16) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (16) | 7 (9)
Gastroenteritis (Infections and infestations) | 4 (7) | 7 (7)
Nasopharyngitis (Infections and infestations) | 55 (74) | 40 (60)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Headache (Nervous system disorders) | 8 (10) | 6 (6)
Hypertension (Vascular disorders) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk Trial Manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.